CLINICAL TRIAL: NCT02491398
Title: Observational Study to Assess the Efficacy and Safety of Bendamustine Plus Rituximab in Patients Affected by Chronic Lymphocytic Leukemia
Brief Title: Efficacy and Safety of Bendamustine Plus Rituximab in Chronic Lympocytic Leukemia
Acronym: LLC1315
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: LLC1315
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- First-line: Previously untreated CLL requiring therapy according to the NCI criteria and treated with at least one cycle of BR as first-line treatment.
  Interventions: Drug: Bendamustine + Rituximab
- Second-line: CLL that received one previous line of treatment using alkylating agents and/or purine analogues with or without monoclonal antibodies, requiring second-line therapy according to the NCI criteria and treated with at least one cycle of BR.
  Interventions: Drug: Bendamustine + Rituximab

INTERVENTIONS:
Drug: Bendamustine + Rituximab

SUMMARY:
This study is intended for Chronic Lymphocytic Leukemia patients who have already undergone a first or second treatment with drugs named bendamustine and rituximab. It will observe the results of this treatment and evaluate its efficacy and side effects.

DETAILED DESCRIPTION:
This cohort study will recruit chronic lymphocytic leukemia (CLL) patients who were treated with first and second-line Bendamustine plus Rituximab (BR) from January 2008 to December 2014 from European centres adhering to the GIMEMA group and the ERIC group, and aims at observing the progression-free survival in CLL patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL / Small Lymphocytic Lymphoma (CLL/) according to the World Health Organisation (WHO) classification 2008.
* Patients who were treated with first and second-line Bendamustine plus Rituximab (BR) from January 2008 to December 2014 from European centres adhering to the GIMEMA group and the ERIC group.
* Previously untreated CLL patients requiring therapy according to the NCI criteria (Hallek M et al, Blood 2008 - Appendix G) and treated with at least one cycle of BR as first-line treatment.
* CLL patients that received one previous line of treatment using alkylating agents and/or purine analogues with or without monoclonal antibodies, requiring second-line therapy according to the NCI criteria (Hallek M et al, Blood 2008 - Appendix G) and treated with at least one cycle of bendamustine and rituximab.
* Age ≥ 18 years old.
* Signed written informed consent according to ICH/EU/GCP and national local law.

Exclusion Criteria:

* Patients who have received 2 or more lines of prior therapy.
* Patients with:

Transformation of CLL into aggressive lymphomas (Richter's Syndrome). HIV infection. Active and uncontrolled HCV and/or HBV infections or liver cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This cohort study will recruit chronic lymphocytic leukemia (CLL) patients who were treated with first and second-line Bendamustine plus Rituximab (BR) from January 2008 to December 2014 from European centres adhering to the GIMEMA group and the ERIC group.
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of patients alive without progression | At 12 months from treatment start
  Progression-free survival

SECONDARY OUTCOMES:
Number of patients untreated | At 12 months from treatment start
  Time-to-next treatment
Number of patients attaining Complete Response (CR) | At six months, that is, at the end of the induction therapy.
Number of patients attainint CR/partial response (PR) | At six months, that is, at the end of the induction therapy.
Number of patients alive | At 12 months from treatment start
Number of patients with grade 3-4 adverse events | At 12 months from treatment start

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cuneo, Study Chair — Ematologia; Azienda Ospedaliera di Ferrara; Gian Matteo Rigolin, Study Director — Ematologia; Azienda Ospedaliera di Ferrara
Locations (41):
- Italy (41):
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. LANCISI - G. SALESI, Ancona
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - S.O.C. di Medicina Interna B - Ospedale - Cardinal Massaia di Asti, Asti
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - Comprensorio Sanitario di Bolzano - Azienda Sanitaria dell'Alto Adige - Ematologia e Centro TMO - Ospedale S.Maurizio, Bolzano
  - ASL N.8 - Ospedale "A. Businco" - Struttura Complessa di Ematologia e CTMO, Cagliari
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - U.O. Ematologia - P.O. Annunziata - A.O. di Cosenza, Cosenza
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - Sez.Ematologia e Dip. scienze Biomediche Arcispedale S. Anna, Ferrara
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - UOC di Ematologia con trapianto Ospedale S. Maria Gorett, Latina
  - Istituto Scientifico Romagnoli per lo Studio e la Cura dei Tumori- IRST, Meldola
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte" P.O. Papardo, Messina
  - Ospedale Niguarda " Ca Granda" - SC Ematologia Blocco SUD, Ponti Est, Scala E, 4° piano, Milan
  - U.O. Ematologia e Trapianto di MIdollo - Ist.Scientifico Ospedale San Raffaele, Milan
  - Unità Trapianto di Midollo Ist. Nazionale Tumori, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Università degli Studi di Padova - Ematologia ed Immunologia Clinica, Padua
  - U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Pagani
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Università di Pisa - Azienda Ospedaliera Pisana - Dipartimento di Oncologia, dei Trapianti e delle nuove Tecnologie in Medicina - Divisione di Ematologia, Pisa
  - Ematologia - Ospedale San Carlo, Potenza
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale "Infermi", Rimini
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Università degli Studi - Policlinico di Tor Vergata, Roma
  - U.O.C. Ematologia e Trapianti - A.O. Senese - Policlinico " Le Scotte", Siena
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari Azienda Ospedaliero-Universitaria, Udine, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - ULSS N.6 Osp. S. Bortolo, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it